CLINICAL TRIAL: NCT05175456
Title: Bed Cooling System to Effect Better Sleep
Brief Title: Use of a Sleep System to Improve Sleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Fitbit LLC (Industry)
Responsible Party: Principal Investigator, Steven Bird, Professor, University of Massachusetts, Worcester
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: H00023479
Record Dates: First submitted 2021-12-14; First posted 2022-01-03 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-02

CONDITIONS: Sleep

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bedjet arm (Experimental): All participants will complete a baseline study period of 4 weeks and then will be provided the Bedjet system.
  Interventions: Other: Bedjet; Device: FitBit

INTERVENTIONS:
Other: Bedjet — Bedjet is a sleep cooling system. All participants will be provided a Bedjet system as part of the study.
Device: FitBit — Each participant will receive a FitBit device to track sleep quality and related information.

SUMMARY:
The purpose of this study is to determine the effect of a bed cooling system on subjective and objective measures of sleep in physicians who work rotating shifts. The intent of the Investigators is to perform a before-and-after trial of a bed cooling system and determine the effects of that cooling system on sleep.

DETAILED DESCRIPTION:
All practicing providers (residents, APPs, and attendings) in the Departments/Divisions of emergency medicine, Ob/Gyn, hospital medicine and family medicine will be offered participation in the study via an email invitation.

Participants will be given a Fitbit device that measures the time of sleep and stages of sleep. Data from the Fitbit are synced to the participant's smart phone. Participants will complete the Single-Quality of Sleep (SQS) scale questionnaire on a daily basis. This questionnaire will be sent to participants on a daily basis via email. This questionnaire is a simple 0-10 rating scale of the quality of their sleep. Participants will then receive the Bedjet cooling sleep system and use it for 10 days to become acclimatized to it. Then they will use the Bedjet for 28 more days, while again completing the daily SQS. This is not a randomized trial, but rather a before-and-after trial.

Changes in mean daily sleep score, SQS from control and intervention time periods will be computed. Subjective measures of participant's satisfaction with the Bedjet system will also be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Residents, Fellows, Clinical Faculty and Advanced Practice Providers (APPs) of UMass Memorial/UMass Medical School who work rotating shifts or nightshifts in Emergency Medicine, Ob/Gyn, Hospital Medicine, or Family Medicine are eligible to participate (pregnant women are also eligible).

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2022-02-05 (Actual); Study Completion 2022-02-05 (Actual)

PRIMARY OUTCOMES:
Sleep Quality Scale change | after 4 weeks
  change in average SQS from before and after time periods Sleep quality information will be evaluated using the Sleep Quality Scale (SQS), an [# of questions] survey that asks questions to obtain information regarding quality of sleep. The range of scores on the survey is [X] to [X], with [X] indicating poor sleep quality and (X] indicating good sleep quality. The outcome will reflect the change in score values from baseline (4 weeks) to post-use of BedJet (4 weeks)
Fitbit Sleep Score | 4 weeks before Bedjet system and the 4 weeks after
  change in average Fitbit Sleep Score from before and after implementation of the Bedjet

CONTACTS AND LOCATIONS:
Locations (1):
- UMassMemorial Health Care, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No